CLINICAL TRIAL: NCT05672953
Title: Biogeography of the Oral Microbiome Using Metatranscriptomic Analyses
Brief Title: Biogeography of the Oral Microbiome
Status: Completed | Type: Observational
Sponsor: Viome (Industry)
Responsible Party: Sponsor
Other Study IDs: V243
Record Dates: First submitted 2022-12-21; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Oral Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study to metatranscriptomically analyze and compare the oral microbiome in different environmental niches within the oral cavity.

DETAILED DESCRIPTION:
This study will collect samples from participants meeting the eligibility criteria over the span of 3 months. Samples will be collected from multiple locations within the oral cavity and metatranscriptomically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older

Exclusion Criteria:

* Positive SARS-CoV-2 test result, if performed
* Antibiotic use in the previous 30 days
* Mouthwash use in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes anyone that meets the inclusion criteria and does not have any exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Species richness in multiple oral locations | 3 months
  Number of species present in different areas swabbed in the oral cavity.

SECONDARY OUTCOMES:
KO richness of multiple oral locations | 3 months
  KO richness of multiple areas swabbed in the oral cavity.

CONTACTS AND LOCATIONS:
Overall Officials: Momchilo Vuyisich, Principal Investigator — Viome; Guruduth Banavar, Principal Investigator — Viome
Locations (1):
- Viome Life Sciences, Bothell, Washington, United States